CLINICAL TRIAL: NCT06795555
Title: Virtual Food for Real Thought: a Pilot Randomised Controlled Trial of Virtual Reality Exposure in Anorexia Nervosa
Brief Title: Virtual Reality Exposure to Reduce Food Related Anxiety in Anorexia Nervosa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Collaborators: University of Salerno, Italy (Unknown); Ospedale S.Bortolo -Vicenza, Italy (Unknown)
Responsible Party: Principal Investigator, CARDI VALENTINA, Associate Professor, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6048/AO/24
Record Dates: First submitted 2025-01-21; First posted 2025-01-28 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Anorexia Nervosa
Keywords: mental health; eating disorders; exposure therapy; virtual reality
MeSH Terms: conditions — Anorexia Nervosa; Psychological Well-Being; Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: Patients are randomly assigned to one of three conditions: (1) treatment as usual + virtual food exposure; (2) treatment as usual + virtual nature exposure; (3) treatment as usual
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Virtual Reality Food Exposure (Experimental): Five sessions of exposure to a virtual kitchen (one session/day, over a week). Participants in this arm will continue receiving treatment as usual for their eating disorder at the treatment center
  Interventions: Behavioral: Virtual reality food exposure
- Virtual Reality Nature Exposure (Active Comparator): Five sessions of exposure to a virtual natural environment (one session/day, over a week). Participants in this arm will continue receiving treatment as usual for their eating disorder at the treatment center
  Interventions: Behavioral: Virtual Reality Nature Exposure
- Treatment as usual (No Intervention): Patients in this condition will receive treatment as usual only

INTERVENTIONS:
Behavioral: Virtual reality food exposure — Patients in this condition are exposed to a virtual kitchen environment once/day, for 5 consecutive days (from Monday, day 1, to Friday, day 5). Each session lasts 5 minutes. The VR environment was specifically developed by the study team (Natali et al, 2024) and it consists of a kitchen with foods of different calorie contents. Patients are invited to explore the environment; they can freely move, open the cupboards and the fridge, and grab and hold the foods. Participants can choose to interact with one of three versions of the virtual kitchen environment: a) a kitchen alone, b) a kitchen with a virtual pet which participants can interact with (and aimed at inducing positive mood) and c) a kitchen with a compassionate avatar which motivates the participant to face food-related fears.
  Arms: Virtual Reality Food Exposure
Behavioral: Virtual Reality Nature Exposure — Patients in this condition complete a session of VR exposure to a natural scenario (from the NatureTreksVR app) for 5 consecutive days (from Monday to Friday), one session/day. Each session lasts 5 minutes. Participants can choose exposure to one of three different natural environments, at the start of each session: a white sand beach ("Blue Ocean"), a snowy mountain ("White Winter"), or a forest in autumn foliage ("Red Fall").
  Arms: Virtual Reality Nature Exposure

SUMMARY:
Exposure to food stimuli often elicit aversive emotions in patients with anorexia nervosa, which can perpetuate eating-related avoidance. Exposure therapy has been shown to effectively reduce anxiety toward, and avoidance of, feared stimuli in several psychiatric disorders. Digital technologies, such as virtual reality (VR) have been employed to implement exposure therapy in situations where in vivo exposure is unfeasible, challenging, or perceived as threatening by patients. VR has also the potential to be used by individuals repeatedly in their own time and environment, to consolidate new learning. This pilot randomised controlled study evaluates the feasibility and clinical impact of repeated VR exposure to food stimuli in patients with anorexia nervosa attending intensive daycare treatment (treatment as usual, TAU). VR food exposure will be compared to the use of a relaxation-focused VR scenario (natural environment) and a control condition (no use of VR). Patients in all groups will receive TAU.

DETAILED DESCRIPTION:
Patients with anorexia nervosa are recruited from daycare services at Eating Disorder Units in Italy. Inclusion criteria are: (1) current diagnosis of anorexia nervosa according to DSM-5 criteria; (2) 14 years or older. Exclusion criteria are: (1) diagnosis of neurological disorders, (2) diagnosis of psychosis or substance abuse disorders, (3) visual/hearing impairments not corrected by glasses/ear implants; (4) non-tolerance of exposure to VR (i.e., cybersickness, dizziness).

Each patient is randomly assigned to one of three conditions: repeated food exposure in a VR kitchen environment + TAU, repeated exposure to a VR natural setting + TAU, or TAU alone .

VR Food Exposure: Patients in this condition undergo one session of VR exposure in a kitchen environment each day for 5 consecutive days (from Monday, day 1, to Friday, day 5). Each session lasts 5 minutes. The VR environment has been specifically developed by the study team and it was tested in a previous one-session study. The scenario consists of a kitchen with foods of different calorie contents either immediately visible in the environment (for example on a table) or stored in drawings, refrigerators, cabinets. Once in the kitchen, patients can freely move, open the cupboards and the fridge, and grab and hold the foods. Patients are invited to explore the environment and interact with the stimuli they feel most comfortable with. Based on their preference, in each session participants access one of three versions of the virtual kitchen: the virtual kitchen alone, a virtual kitchen + a pink elephant (designed to induce positive mood), or a virtual kitchen + a reassuring voice that encourages to interact with foods and face food-related fears.

VR Nature Exposure: Patients in this condition undergo one session of VR exposure to a natural scenario each day, for 5 consecutive days (from Monday to Friday), through the NatureTreks app. Each session lasts 5 minutes. Participants perform the exposure while seated, and are instructed to observe the environment and try to relax. Based on their preference, in each session participants are able to choose one of three different natural environments: a white sand beach ("Blue Ocean"), a snowy mountain ("White Winter"), or a forest in autumn foliage ("Red Fall")

TAU: It consists of a daycare program (attendance Monday to Friday) including individual psychological therapy (based on cognitive-behavioral principles), nutritional counseling, assisted meals, group activities (e.g., psychotherapy, art therapy, music therapy, relaxation protocols), and psychoeducation for family members. For ethical reasons, at the end of the follow-up assessment, participants in the control group are given the opportunity to engage in VR exposure.

Patients in all conditions complete a baseline (day 0) and end of intervention (day 5) assessment. The baseline assessment includes:

* Demographic questionnaire (age, years of education, current pharmacological treatments, height, weight)
* Eating Disorder Examination Questionnaire
* Depression, Anxiety and Stress Scale
* Difficulties in Emotion Regulation Scale
* Positive and Negative Affect Schedule
* State and Trait Anxiety Scale
* Motivational Ruler: patients are asked to rate, on a scale from 0 to 10 importance and ability to change.
* Food evaluation: patients are asked to rate, on a scale from 0 to 100 wanting, liking and fear of 21 foods of different caloric content.
* Meal related anxiety: just before starting their meal at the hospital, patients are asked to rate their current level of anxiety on a scale from 0 to 10.

The PANAS, the STAI, the motivational ruler, food evaluation, and meal related anxiety are completed at the end of intervention.

Each day, immediately before and after the exposure, participants in the food and nature exposure groups are asked to rate, on a scale from 0 to 100, their anxiety in the moment and also the anxiety they feel when thinking of the next meal. At the end of each exposure session, they are asked to rate their sense of presence and discomfort in the VR environment.

ELIGIBILITY:
Inclusion Criteria:

* current diagnosis of anorexia nervosa according to DSM-5 criteria
* 14 years or older.

Exclusion Criteria:

* diagnosis of neurological disorders
* diagnosis of psychosis or substance abuse disorders
* visual/hearing impairments not corrected by glasses/ear implants
* non-tolerance of exposure to VR (i.e., cybersickness, dizziness)

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to end of intervention in meal related anxiety | Measurements at baseline and day 5
  Meal related anxiety is assessed on a Likert scale from 0 (no anxiety) to 10 (extreme anxiety)
Feasibility of exposure to the virtual reality environments | Following each of five exposure sessions, over a time period of five days
  Percentage of participants who interrupt exposure to the virtual reality environment before completion.
  Discomfort associated to the virtual reality exposure session, rated at the end of each session on a visual analogue scale (0-100).

SECONDARY OUTCOMES:
Change from baseline to end of treatment in positive and negative affect | Measurements at baseline and day 5
  The PANAS is a validated self-report instrument consisting of two subscales assessing respectively positive and negative affect. The score of each subscale can range from 10 to 50, with higher scores representing higher levels of positive/negative affect.
Change from baseline to end of intervention in state anxiety | Measurements at baseline and day 5
  The STAI state is a 20-item self-report scale for the assessment of state anxiety. Possible scores range from 0 to 80 and greater scores indicate greater anxiety
Change from baseline to end of intervention in food pictures evaluation | Measurements at baseline and day 5
  Food-related wanting, liking and fear will be measured in response to the presention of 21 pictures of foods of different caloric content, using a scale from 0 (not at all) to 100 (extremely).
Effect sizes of changes in anxiety and meal related anxiety from before to after virtual reality exposure | Measurements before and after each exposure session, over five days
  Ratings of general and meal related anxiety will be collected at the beginning and at the end of each virtual reality exposure session through a visual analogue scale ranging from 0 to 100.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Padova, Padua, Italy, Italy

IPD SHARING:
Plan to Share IPD: No
a plan will be established by the research team for data sharing following publication of the first manuscript

REFERENCES:
- [Background] Gratz, K.L., Roemer, L. Multidimensional Assessment of Emotion Regulation and Dysregulation: Development, Factor Structure, and Initial Validation of the Difficulties in Emotion Regulation Scale. Journal of Psychopathology and Behavioral Assessment 26, 41-54 (2004). https://doi.org/10.1023/B:JOBA.0000007455.08539.94
- [Background] Terracciano A, McCrae RR, Costa PT Jr. Factorial and construct validity of the Italian Positive and Negative Affect Schedule (PANAS). Eur J Psychol Assess. 2003;19(2):131-141. doi: 10.1027//1015-5759.19.2.131. PMID 20467578
- [Background] Bottesi G, Ghisi M, Altoe G, Conforti E, Melli G, Sica C. The Italian version of the Depression Anxiety Stress Scales-21: Factor structure and psychometric properties on community and clinical samples. Compr Psychiatry. 2015 Jul;60:170-81. doi: 10.1016/j.comppsych.2015.04.005. Epub 2015 Apr 15. PMID 25933937
- [Background] Calugi S, Milanese C, Sartirana M, El Ghoch M, Sartori F, Geccherle E, Coppini A, Franchini C, Dalle Grave R. The Eating Disorder Examination Questionnaire: reliability and validity of the Italian version. Eat Weight Disord. 2017 Sep;22(3):509-514. doi: 10.1007/s40519-016-0276-6. Epub 2016 Apr 2. PMID 27039107